CLINICAL TRIAL: NCT02544412
Title: A Well-being Training for Preservice Teachers
Acronym: PST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other); The Trust for the Meditation Process (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-1263; A487400 (Other: UW, Madison); L&S/PSYCHOLOGY/PSYCHOLOGY (Other: UW, Madison)
Record Dates: First submitted 2015-09-02; First posted 2015-09-09 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Burnout, Professional; Stress, Psychological; Well-being; Psychological Adjustment; Self-regulation
Keywords: Mindfulness; School Teachers; preservice teachers; teacher education
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological; Self-Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): A novel mindfulness-based well-being training for preservice teachers will be employed. The intervention will be held once a week for 8-10 weeks. Two 4-hour "days of mindfulness" will also be implemented during the intervention period. The intervention will involve training in a range of attentional and constructive (Dahl, Lutz, & Davidson) contemplative practices. During the follow-up period participants will receive weekly 15 minute "booster" trainings.
  Interventions: Behavioral: novel mindfulness-based well-being training
- Control Group (No Intervention): Teacher education as usual. These participants will continue with the prescribed teacher training regime established by the Early Education Certification Program at the university.

INTERVENTIONS:
Behavioral: novel mindfulness-based well-being training
  Arms: Intervention Group

SUMMARY:
The purpose of this project is to study whether a mindfulness-based training program supports self-regulation, resiliency, effective classroom behaviors, and persistence in teaching.

DETAILED DESCRIPTION:
Participants in this study will be undergraduate pre-service teachers already enrolled in the Early Elementary Certification Program (EECP) in the School of Education. This competitive admission program is four semesters long and consists of 4 certificate granting areas. Over the course of 2 years (i.e., 4 semesters), the investigators will recruit a total of 8 cohorts; 2 from each certificate granting area. Participants will be recruited during their second semester in the program for enrollment during the third semester (i.e., enrollment first semester of senior year). Cohorts will be match randomized by cohort type, ensuring that 4 cohorts are randomized to treatment and 4 cohorts are randomized to teacher education as usual, and that one of each type of cohort is randomized to treatment and control, respectively.

All participants will complete a battery of self-report and behavioral tasks, as well as undergo a standardized classroom observation prior to the start of the intervention, immediately after the intervention, and at follow-up (5-8 months post intervention). Follow-up testing will occur during the final month of the final semester in the EECP program, a time during which participants will be full-time student teaching, training that best approximates in-service teaching. The qualitative component of this study will involve participants partaking in approximately four-hours of interviews (either group or individual based on a hierarchal sampling criterion), before and after the intervention period. In addition, all student EECP records will be qualitatively analyzed (i.e., supervisor notes, state certification portfolios). Each September for three years post-graduation, participants will be contacted and instructed to complete an online survey consisting of self-report inventories and information about whether they are continuing to teach and if so, the name and district of the school they currently work.

Participants randomized to treatment will receive 1.5 hours of mindfulness training for 8 to 10 weeks during their third semester. Thirty minutes of this will occur during mandatory cohort seminar time, with the remaining one-hour after the end of cohort seminar time. In addition, during the intervention period they will participate in two 4-hour "Days of Mindfulness." In total, intervention participants will receive about 21 hours of instruction in mindfulness over the intervention period. During the following semester (4th semester), intervention participants will receive 15 minutes of mindfulness "booster" practice each week as part of their mandatory cohort seminar.

This novel mindfulness based intervention is incorporates elements of Mindfulness Based Stress Reduction (Kabat-Zinn, 1982), as well as contemplative practices that might be defined as social connectedness practices or constructivist practices (Dahl, Lutz, & Davidson, 2015). The curriculum has been developed by experienced mindfulness teachers (>10 years teaching experience, on average), all of whom have extensive meditation histories and most of whom have long-term experience as classroom teachers. The training will consist of formal and informal mindfulness meditation practices.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students in good academic standing entering their third semester of one of the following teacher education certificate programs (Early Education ESL, Middle Education SPED, Middle Education Content, Middle Education ESL). Note that good academic standing is a requirement for continuation in the certification program.

Exclusion Criteria:

* A history of schizophrenia-spectrum, bipolar disorder, or other psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline on CLASS assessment tool (La Paro, Pianta, & Stuhlman, 2004) | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  A standardized classroom observation tool assessing teacher classroom behaviors.
Change from baseline on Symptoms Checklist 90 Revised (Derogatis, 1994) | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  a 90-item self-report of psychological symptoms comprised of 9 symptom axes (somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism). An aggregated score across all 9 domains provides a Global Severity Index score of psychological health.
Change from baseline on Maslach Burnout Inventory - Education Survey (Maslach, Jackson, & Leiter, 1996) | 1-2 weeks before intervention (i.e., baseline), 11-12 weeks after baseline (1-2 weeks post-intervention), 8-11 months after baseline (5-8 months post-intervention): ~14 months after baseline, ~26 months after baseline, and ~38 months after baseline
  a 22-item self-report of teaching related burnout
Change from baseline on Emotional go/nogo (Hare et al., 2008) | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  An emotional inhibition paradigm.
Persistence in teaching: Current profession and role (if teaching, name of school) | ~ 14 months after baseline, ~ 26 months after baseline, and ~ 38 months after baseline.
  Self-report on employment status following graduation and teacher licensure.

SECONDARY OUTCOMES:
Change from baseline on Implicit Positive and Negative Affect Test (Quirin, Kazen, & Kuhl, 2009) | 1-2 weeks before intervention (i.e., baseline), 11-12 weeks after baseline (1-2 weeks post-intervention), 8-11 months after baseline (5-8 months post-intervention): ~14 months after baseline, ~26 months after baseline, and ~38 months after baseline
  A computer-based behavioral measure of implicit affective bias in which participants are provided with 5 nonsense words and asked to rate the words on a scale of emotional valence.
Change from baseline on General Self-efficacy Scale (Jerusalem & Schwarzer, 1992) | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  A 10-item self-report of general self-efficacy
Change from baseline on Psychological Well-Being Scale (Ryff & Keyes, 1995) | 1-2 weeks before intervention (i.e., baseline), 11-12 weeks after baseline (1-2 weeks post-intervention), 8-11 months after baseline (5-8 months post-intervention): ~14 months after baseline, ~26 months after baseline, and ~38 months after baseline
  A 54-item self-report inventory assessing psychological well-being.
Change from baseline on Positive and Negative Affect Schedule (Watson, Clark, & Tellegen, 1988) | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  A self-report survey of general positive and negative affect.
Change from baseline on Emotional Styles Questionnaire (under development) | 1-2 weeks before intervention (i.e., baseline), 11-12 weeks after baseline (1-2 weeks post-intervention), 8-11 months after baseline (5-8 months post-intervention): ~14 months after baseline, ~26 months after baseline, and ~38 months after baseline
  A self-report designed to assess styles of emotional responding.
Change from baseline on Open response on difficulties in teaching | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  A one-item open response on difficulty in teaching.
Change from baseline on Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983) | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  A 10-item self-report on perceived stress in the last month.
Change from baseline on Implicit Association Task (Race, child and adult versions; Baron & Banaji, 2006) | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  A behavioral task designed to assess implicit biases related to race.
Change from baseline on Five Facet Mindfulness Questionnaire (Baer et al., 2008) | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  A 39-item self-report of mindfulness
Change from baseline on Breath Count Task (Levinson et al., 2014) | 1-2 weeks before intervention (i.e., baseline), 11 - 12 weeks after baseline (1-2 weeks post-intervention), 8 - 11 months after baseline ( 5-8 months post intervention)
  15 minute behavioral measure of mindfulness

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flook, PhD, Principal Investigator — University of Wisconsin, Madison; Matthew J Hirshberg, PhD, Study Director — University of Wisconsin, Madison
Locations (1):
- UW Madison Department of Curriculum and Instruction, Madison, Wisconsin, United States

REFERENCES:
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] La Paro, K. M., Pianta, R. C., & Stuhlman, M. (2004). The Classroom Assessment Scoring System: Findings from the prekindergarten year. The Elementary School Journal, 104(5), 409-426. http://doi.org/10.1086/499760
- [Background] Levinson DB, Stoll EL, Kindy SD, Merry HL, Davidson RJ. A mind you can count on: validating breath counting as a behavioral measure of mindfulness. Front Psychol. 2014 Oct 24;5:1202. doi: 10.3389/fpsyg.2014.01202. eCollection 2014. PMID 25386148
- [Background] Dahl CJ, Lutz A, Davidson RJ. Reconstructing and deconstructing the self: cognitive mechanisms in meditation practice. Trends Cogn Sci. 2015 Sep;19(9):515-23. doi: 10.1016/j.tics.2015.07.001. Epub 2015 Jul 28. PMID 26231761
- [Background] Derogatis, L. R. (1994). SCL-90-R Symptom Checklist-90-R administration, scoring and procedures manual. Minneapolis, MN: National Computer Systems.
- [Background] Maslach, C., Jackson, S. E., & Leiter, M. P. (1996). Maslach burnout inventory manual . Mountain View, CA: CPP. Inc., and Davies-Black.
- [Background] Baron AS, Banaji MR. The development of implicit attitudes. Evidence of race evaluations from ages 6 and 10 and adulthood. Psychol Sci. 2006 Jan;17(1):53-8. doi: 10.1111/j.1467-9280.2005.01664.x. PMID 16371144
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Quirin M, Kazen M, Kuhl J. When nonsense sounds happy or helpless: The Implicit Positive and Negative Affect Test (IPANAT). J Pers Soc Psychol. 2009 Sep;97(3):500-16. doi: 10.1037/a0016063. PMID 19686004
- [Background] Jerusalem, M., & Schwarzer, R. (1992). Self-efficacy as a resource factor in stress appraisal processes. Self-efficacy: Thought control of action, 195-213.
- [Background] Ryff CD, Keyes CL. The structure of psychological well-being revisited. J Pers Soc Psychol. 1995 Oct;69(4):719-27. doi: 10.1037//0022-3514.69.4.719. PMID 7473027
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Hare TA, Tottenham N, Galvan A, Voss HU, Glover GH, Casey BJ. Biological substrates of emotional reactivity and regulation in adolescence during an emotional go-nogo task. Biol Psychiatry. 2008 May 15;63(10):927-34. doi: 10.1016/j.biopsych.2008.03.015. PMID 18452757